CLINICAL TRIAL: NCT00273572
Title: The Effect of a Lifestyle Intervention Program on Parameters of the Metabolic Syndrome Among Non-Diabetic Obese Arab Women
Brief Title: Lifestyle Intervention in Obese Arab Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: D-Cure, Israel (Industry); Chief Scientist, The Israel Ministry of Science (Unknown)
Responsible Party: Ofra Kalter, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-04-3335-OK-CTIL
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Metabolic Syndrome; Diabetes
Keywords: Obesity; Women; Arab; Metabolic syndrome; Lifestyle intervention; Quality of life
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate lifestyle intervention (Active Comparator): Moderate lifestyle intervention including two group sessions and one individual counselling session with a nutritionist, at recruitment. Individual sessions with a nutritionist after 6 and 12 months on follow-up.
  Interventions: Other: Moderate Lifestyle Intervention
- Intensive lifestyle intervention (Experimental): Intensive lifestyle intervention, including bi-monthly group sessions with a physical activity instructor; a monthly group session with a nutritionist, and a monthly individual session with a nutritionist.
  Interventions: Other: Intensive lifestyle intervention

INTERVENTIONS:
Other: Moderate Lifestyle Intervention — Two educational group meetings with a dietitian in the first month of intervention; One individual counselling session with a dietitian at baseline, and at 6-month and 12-month follow-up
  Other Names: Lifestyle intervention
  Arms: Moderate lifestyle intervention
Other: Intensive lifestyle intervention — A monthly individual counselling session with a dietitian; A monthly group session with a dietitian; Bi-monthly group sessions with a physical activity instructor
  Other Names: Lifestyle intervention
  Arms: Intensive lifestyle intervention

SUMMARY:
The study protocol aims to test the hypothesis that a lifestyle intervention program aimed to increase leisure-time physical activity and reduce body weight will improve the parameters of the metabolic syndrome and quality of life among obese, non-diabetic Arab women

DETAILED DESCRIPTION:
200 obese non-diabetic Arab women, 35-54 years old, with one or more parameters of the metabolic syndrome (NCEP-III criteria) will be randomized to either conventional or intensive treatment. The intensive intervention arm will include group meetings with physical education instructor (twice a month),group meetings with a dietician (once per month) and personal dietary counselling (once per month). The targets to be achieved will be at least 7% reduction of the initial body weight and engagement in leisure-time sports activity for at least 150 min/week.Evaluation before enrollment and at the end of the trial will include: information on dietary and physical activity habits, quality of life parameters, anthropometric and blood pressure measurement, blood lipid profile, and fasting and post oral glucose load blood glucose and insulin levels. Duration of the intervention: 12 month.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI: 30-40 kg/squared meter)
* Female Gender
* Being 35-54 years old

Exclusion Criteria:

* Diabetic

A contraindication for physical activity

Ages: 35 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2004-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Parameters of the metabolic syndrome | At baseline, and after 6 and 12 months

SECONDARY OUTCOMES:
Quality of life | At baseline, and after 12 months
Attainment of weight reduction and physical activity targets | At baseline, and after 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Kalter - Leibovici, M.D., Principal Investigator — Director, Unit of Cardiovascular Epidemiology, Gertner Institute for Epidemiology & Health Policy Research, Sheba Medical Center, ISRAEL
Locations (1):
- Unit of Cardiovascular Epidemiology, Gertner Institute for Epidemiology & Health Policy Research, Sheba Medical Center, Tel-Hashomer, Ramat-Gan, Israel

REFERENCES:
- [Derived] Kalter-Leibovici O, Younis-Zeidan N, Atamna A, Lubin F, Alpert G, Chetrit A, Novikov I, Daoud N, Freedman LS. Lifestyle intervention in obese Arab women: a randomized controlled trial. Arch Intern Med. 2010 Jun 14;170(11):970-6. doi: 10.1001/archinternmed.2010.103. PMID 20548010